CLINICAL TRIAL: NCT03030781
Title: Relationship of Cricoid With the Right and Left Bronchial Diameters in the Pediatric Population Using Three-dimensional Imaging.
Status: Completed | Type: Observational
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Tariq Wani, CONSULTANT ANESTHESIOLOGIST, King Fahad Medical City
Other Study IDs: H-01-R-012, 17-010
Record Dates: First submitted 2017-01-21; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-11

CONDITIONS: Larynx; Oxygen; Intubation
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Specific and objective guidelines for choosing endobronchial tube size for main-stem intubation in pediatric patients are lacking. The objective criteria for choosing an ETT size for OLV are likely to increase the safety and success. The primary aims of this study were to define the relationship between cricoid and mainstem bronchi (right and left) in children of various ages and to determine the effects of age, height and weight.

DETAILED DESCRIPTION:
Understanding the relationship between cricoid and mainstem bronchi can provide to be a useful adjunct for lung isolation in children. The relationship between cricoid dimensions and the dimensions of main-stem bronchi (right and left) have been studied using 2 dimensional CT images and video-bronchoscopic images. The present study defines the volume-based relationship between the right main-stem bronchus (RMSB), left main-stem bronchus (LMSB) and the cricoid ring based on 3 dimensional CT derived images.

Methods: The three dimensional CT images of 35 children, younger than 8 years, undergoing radiological evaluation unrelated to airway symptomatology were examined. The children were evaluated during spontaneous ventilation without airway devices either during natural sleep or with sedation. The 3-dimensional images of the airway column were evaluated at the level of cricoid, right mainstem bronchus and left main-stem bronchus, volumes were calculated and comparisons made between these levels. Univariate and multivariate regression analysis was used to determine whether one or more of the variables (age, gender, height, weight and cricoid) had a predictable relationship to the RMSB and the LMSB diameter.

ELIGIBILITY:
Inclusion Criteria:

* Children 1 month to 8 years of age

Exclusion Criteria:

* Patients with tracheostomy Tracheoesophageal fistula Presence of mediastinal mass Diaphragmatic hernia Preterm infants

Ages: 1 Month to 96 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The present study evaluated CT images of the chest of children less than 8 years of age. The database search of the electronic medical records identified 110 patients of which 40 patients qualified for the study.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
comparison between cricoid and mainstem borncchi | 1 month to 8 years

IPD SHARING:
Plan to Share IPD: No